CLINICAL TRIAL: NCT06875401
Title: Long-Term Patient-Reported Maternal Outcomes Following Abdominal Cerclage for the Prevention of Preterm Birth
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-45-70-80-24
Record Dates: First submitted 2025-03-06; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Cerclage, Cervical; Cervical Insufficiency
Keywords: Patient reported outcomes (PRO); Quality of life; Preterm birth; Abdominal cerclage
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Transabdominal cerclage: Participants with a transabdominal cerclage and subsequent birth
  Interventions: Procedure: Abdominal cerclage (open or laparoscopic)
- No abdominal cerclage, CS: Participants with no abdominal cerclage, but previous caesarean section. Participants matched on birth mode and -year, and age at time of cohort entry.
- No abdominal cerclage, vaginal birth: Participants matched on birth year and age at time of cohort entry. Participants with a history of C-section and/or instrumental deliveries cannot enter this comparison group.
- Women with a transabdominal cerclage and no subsequent birth: Participants who underwent the abdominal cerclage procedure, but did not become pregnant after the procedure.
  Interventions: Procedure: Abdominal cerclage (open or laparoscopic)

INTERVENTIONS:
Procedure: Abdominal cerclage (open or laparoscopic) — Participants who have had either an open transabdominal cerclage or laparoscopic abdominal cerclage procedure performed.
  Groups: Transabdominal cerclage; Women with a transabdominal cerclage and no subsequent birth

SUMMARY:
This study aims to explore the maternal patient reported outcomes on pelvic pain sexual health anxiety and depression bladder discomfort foreign body sensation trust in the cerclage, and how these parameters affect the general health perception in the quality of life of women treated with abdominal cerclages in Denmark since 2004.

ELIGIBILITY:
Inclusion Criteria:

* Transabdominal cerclage

Exclusion Criteria:

* Most recent birth within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female biological sex
Study Population: 1. Participants with a TAC compared to controls with no TAC.
  2. Participants exposed to short versus longer time spans since TAC insertion.
  3. Participants with a TAC and no subsequent birth versus TAC and at least one subsequent birth.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
General Health Perception scale - SF-36 | At enrollment
  The difference in general health perception as measured by patient reported outcome measures (PROMS) in participants treated with TAC. A difference of 10 points or more is regarded as a clinically relevant difference.
Hospital anxiety and depressen scale (HADS) | At enrollment
  The difference in depression and anxiety scores as measured by PROMS in participants who did not give birth since the TAC. The outcome is categorized in normal, borderline abnormal or abnormal.

SECONDARY OUTCOMES:
Pelvic pain | At enrollment
  This issue was conceptualized as pelvic or vaginal pain (pressure, sharp, cramping or pulling) that may be intermittent and worsens with activity or at the end of the day.
  Questionnaire: The Danish Chronic Pelvic Pain Questionnaire
Foreign body sensation | At enrollment
  This issue was conceptualized as awareness and reminding of having the cerclage. Consists of two qualitatively pilot tested ad hoc questions.
Trust in the cerclage | At enrollment
  This issue was conceptualized as trust in the effectiveness of the cerclage to prevent preterm birth. Consists of two qualitatively pilot tested ad hoc questions.
Bladder discomfort | At enrollment
  This issue was conceptualized bladder discomfort as "Frequency, nocturia, urgency, urge incontinence (overactive bladder), Incontinence, bladder pain". The Bristol Female Lower Urinary Tract Symptoms questionnaire - short form (ICIQ-FLUTS-SF).
  * Filling (4 items, maximum score 16)
  * Voiding (3 items, maximum score 12)
  * Incontinence (4 items, maximum score 16)
Sexual health | At enrollment
  This issue was conceptualized as sexual desire, arousal and dyspareunia. Questionnaire: Female Sexual Function Index Scoring (FSFI).
  * Desire (2 items, maximum score 6)
  * Arousal (4 items, maximum score 6)
  * Lubrication (4 items, maximum score 6)
  * Orgasm (3 items, maximum score 6)
  * Satisfaction (3 items, maximum score 6)
  * Pain (3 items, maximum score 6)
SF - 36 QOL | At enrollment
  * Physical functioning (10 items, maximum score 100)
  * Role limitations due to physical health problems (4 items, maximum score 100)
  * Role limitations due to emotional problems (3 items, maximum score 100)
  * Energy/fatigue (4 items, maximum score 100)
  * Emotional well-being (5 items, maximum score 100)
  * Social functioning (2 items, maximum score 100)
  * Bodily pain (2 items, maximum score 100)
  * General health perceptions (5 items, maximum score 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided